CLINICAL TRIAL: NCT04867044
Title: Prevalence of Temporomandibular Disorders in Patients With Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Yerkoy State Hospital (Other)
Responsible Party: Principal Investigator, Başak Çiğdem Karaçay, Spesialist, Yerkoy State Hospital
Other Study IDs: 2017-KAEK-189_2021.03.10_17
Record Dates: First submitted 2021-04-22; First posted 2021-04-30 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Temporomandibular Disorder; Fibromyalgia
Keywords: fibromiyalgia syndrome; Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STUDY GROUP: patient diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria
  Interventions: Other: STUDY
- CONTROL GROUP: healthy women volunteers
  Interventions: Other: Control

INTERVENTIONS:
Other: STUDY — One Hundred Fifty woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria
  Other Names: Fibromiyalgia Patient
  Groups: STUDY GROUP
Other: Control — healthy woman volunteers
  Other Names: healthy participant
  Groups: CONTROL GROUP

SUMMARY:
One Hundred Fifty woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria and 150 healthy woman volunteers will be included.Demographic data (age, gender, height, weight, marital status, education level) and duration of fibromyalgia diagnosis will be recorded. Patients will be evaluated according to the Diagnostic Criteria for Temporomandibular Disorders: Assessment Instruments (DCTMD: AI ). Patients will be evaluated by Diagnostic Criteria for Temporomandibular Disorders: Temporomandibular Disorders (TMD) Pain Screener, Symptom questionnaire, Clinical Examination Form from Assessment Instruments Axis I. Pain Drawing, Graded Chronic Pain (version 2), Jaw Functional Limitation Scale-8 (JFLS-8), Patient Health Questionnaire (PHQ-4), Oral Behaviors Checklist will be applied within the scope of Axis II.

DETAILED DESCRIPTION:
In our study, the investigators aim to compare the frequency of temporomandibular disorders between healthy female participants and female patients diagnosed with fibromyalgia.

Our study will consists of 300 female participants aged between 18 and 65 years who applied to the physical therapy and rehabilitation outpatient clinic between May 2021 and August 2021. This case-control study will conducted according to the Declaration of Helsinki. Participants gave written voluntary consent and enrolled in this case-control study. One Hundred Fifty woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria and 150 healthy woman volunteers will be included. Patients with temporomandibular region surgery, congenital teporomandibular joint pathologies, and previous temporomandibular region trauma were will be excluded from the study. Because fibromyalgia is a disease that mostly affects women, the investigators designed our study so that all participants were women. In addition, demographic data (age, gender, height, weight, marital status, education level) and duration of fibromyalgia diagnosis will be recorded. Patients will be evaluated according to the Diagnostic Criteria for Temporomandibular Disorders: Assessment Instruments ( DCTMD: AI ). Patients will be evaluated by Diagnostic Criteria for Temporomandibular Disorders: TMD Pain Screener, Symptom questionnaire, Clinical Examination Form from Assessment Instruments Axis I. Pain Drawing, Graded Chronic Pain (version 2), Jaw Functional Limitation Scale-8 (JFLS-8), Patient Health Questionnaire (PHQ-4),Oral Behaviors Checklist will be applied within the scope of Axis II.

ELIGIBILITY:
Inclusion Criteria:

* One hundred fifty woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria
* One hundred fifty womanhealthy volunteers

Exclusion Criteria:

* Patients with temporomandibular region surgery
* Congenital teporomandibular joint pathologies
* Previous temporomandibular region trauma were excluded from the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Our study consists of 300 female participants aged between 18 and 65 years
Study Population: Our study consists of 300 female participants aged between 18 and 65 years who applied to the physical therapy and rehabilitation outpatient clinic.. One Hundred Fifty woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria and 150 healthy woman volunteers were included.Because fibromyalgia is a disease that mostly affects women, we designed our study so that all participants were women.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
DCTMD: AI Axis I Pain Screener | 0 DAY
  TMD Pain Screener which is a simple, reliable, and valid self-report instrument used to assess for the presence of any pain-related TMD, with sensitivity and specificity ≥ 0.95 which is recommended for all patients in any clinical setting. A positive screen is followed by further evaluation to arrive at the specific TMD pain-related diagnoses.
DCTMD: AI Axis I Symptom questionnaire | 0 DAY
  Symptom questionnaire which assess pain characteristics as well as history of jaw noise, jaw locking, and headache.
DCTMD: AI Axis I Clinical Examination Form | 0 DAY
  Clinical Examination Form- The clinical examination includes provocation tests for TMJ arthralgia of pain with any jaw movement (ie, opening, lateral, and protrusive) and TMJ palpation. For myalgia, the tests include pain with opening jaw movements and palpation of the temporalis and masseter muscles.

SECONDARY OUTCOMES:
DCTMD: AI Axis II-Pain Drawing | 0 DAY
  Pain Drawing-pain drawing of the head, jaw, and body, and it allows the patient to report the location of all pain complaints
DCTMD: AI Axis II-Graded Chronic Pain (version 2) | 0 DAY
  Graded Chronic Pain (version 2) is a short, reliable, and valid instrument that assesses pain intensity and pain-related disability.10 The two GCPS subscales are: Characteristic Pain Intensity (CPI), which reliably measures pain intensity, with ≥ 50/100 considered "high intensity," and the pain-disability rating, which is based on number of days that pain interferes with activity and on extent of interference with social, work, or usual daily activities
DCTMD: AI Axis II-Jaw Functional Limitation Scale-8 (JFLS-8) | 0 DAY
  Jaw Functional Limitation Scale-8 (JFLS-8) which assesses global limitations across mastication, jaw mobility, and verbal and emotional expression
DCTMD: AI Axis II-Patient Health Questionnaire (PHQ-4) | 0 DAY
  Patient Health Questionnaire (PHQ-4) is a short, reliable, and valid screening instrument for detecting "psychological distress" due to anxiety and/or depression in patients in any clinical setting.A cutoff of > 6, suggesting moderate psychological stress, should be interpreted as warranting observation, while a cutoff of > 9, suggesting severe psychological distress, should be interpreted as warranting either further assessment or referral
DCTMD: AI Axis II- Oral Behaviors Checklist (OBC) | 0 DAY
  Oral Behaviors Checklist (OBC), which assesses the frequency of oral parafunctional behaviors.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Basak Cigdem karacay, Yozgat, Yerkoy
  - Basak CigdemKaracay, Yozgat, Yerkoy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moreno-Fernandez AM, Jimenez-Castellanos E, Iglesias-Linares A, Bueso-Madrid D, Fernandez-Rodriguez A, de Miguel M. Fibromyalgia syndrome and temporomandibular disorders with muscular pain. A review. Mod Rheumatol. 2017 Mar;27(2):210-216. doi: 10.1080/14397595.2016.1221788. Epub 2017 Feb 1. PMID 27539739
- [Background] Fujarra FJ, Kaziyama HH, Siqueira SR, Yeng LT, Camparis CM, Teixeira MJ, Siqueira JT. Temporomandibular disorders in fibromyalgia patients: are there different pain onset? Arq Neuropsiquiatr. 2016 Mar;74(3):195-200. doi: 10.1590/0004-282X20160017. PMID 27050847
- [Background] Pimentel MJ, Gui MS, Martins de Aquino LM, Rizzatti-Barbosa CM. Features of temporomandibular disorders in fibromyalgia syndrome. Cranio. 2013 Jan;31(1):40-5. doi: 10.1179/crn.2013.006. PMID 23461261